CLINICAL TRIAL: NCT01611012
Title: The Development of a Clinical Test to Assess the Inflammatory Phenotype of Asthma
Acronym: AIR
Status: Completed | Type: Observational
Sponsor: Prof. Jan-Willem Lammers MD PhD (Other)
Responsible Party: Sponsor-Investigator, Prof. Jan-Willem Lammers MD PhD, M.D. PhD, UMC Utrecht
Organization: UMC Utrecht (Other)
Other Study IDs: AIR2012
Record Dates: First submitted 2012-05-25; First posted 2012-06-04 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
Keywords: Asthma; Inflammation; Phenotype; Sputum
MeSH Terms: conditions — Asthma; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Leukocytes in peripheral blood, serum samples for protein profiling and sputum samples.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the type and degree of inflammatory parameters in peripheral blood of asthma patients compared to analysis of induced sputum.

115 asthma patients visiting the outpatient clinic of the University Medical Center will be included. Blood samples are obtained and sputum induction is performed.

Hypothesis: in asthma the analysis of type and degree of inflammation in peripheral blood by changes in phenotypes of leukocytes is at least as reliable as analysis of cells obtained from induced sputum

DETAILED DESCRIPTION:
Asthma is a heterogeneous disease and can be classified by level of control, disease severity and the inflammatory phenotype. However, these different domains overlap and classification of patients according to these characteristics has caused confusion in the literature. Concerning the inflammatory phenotype international consensus is present regarding the diagnostic power of induced sputum. This methodology is, however, difficult to implement in general practice. Local inflammation is associated with a complex combination of systemic pro- and anti-inflammatory signals that induce changes in responsive leukocytes. These changes can be used as read-out for type and degree of inflammatory disease. Hypothesis: This will facilitate the diagnosis of inflammatory phenotypes in asthma, as general application of induced sputum is not feasible.

Goals

1. To investigate whether analysis of antibodies directed against active Beta-1 and Beta-2-integrins (CD29/CD18) and FcγRII (CD32) of primed eosinophils allows the diagnosis of eosinophilic asthma as compared to analysis of sputum eosinophilia.
2. To evaluate the applicability of antibodies against active β1/β2-integrins and FcγRII in symptomatic asthma patients as a test to diagnose eosinophilic and neutrophilic asthma.
3. To determine specific protein profiles in serum of asthma patients by proteomics for the development of a diagnostic test.
4. To evaluate the effectiveness of this new test in comparison with FeNO.

ELIGIBILITY:
Inclusion Criteria:

* Adult asthma
* Aged 18-75 years
* Visiting the outpatient clinic of the UMCU

Exclusion Criteria:

* Smoking at present or in the last 12 months
* Past smoking history of > 10 Pack years
* AB treatment for RTI in past 4 weeks
* ABPA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma patients between the age of 18 and 75, visiting outpatient respiratory clinic of the University Medical Centre in Utrecht, The Neterlands.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
inflammatory phenotype | 1 day
  inflammatory phenotype in blood compared to type in sputum

SECONDARY OUTCOMES:
Measurement of antibodies against active β1/β2-integrins and FcγRII | 1 day
Measuring specific protein profiles in serum of asthma patients by proteomics | 1 day
FENO | 1 day
  Fraction of Exhaled Nitric Oxide

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Willem Lammers, MD, PhD, Principal Investigator — Respiratory Department, UMC Utrecht; Leo Koenderman, M.D. PhD, Study Chair — Respiratory Department, UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Kanters D, ten Hove W, Luijk B, van Aalst C, Schweizer RC, Lammers JW, Leufkens HG, Raaijmakers JA, Bracke M, Koenderman L. Expression of activated Fc gamma RII discriminates between multiple granulocyte-priming phenotypes in peripheral blood of allergic asthmatic subjects. J Allergy Clin Immunol. 2007 Nov;120(5):1073-81. doi: 10.1016/j.jaci.2007.06.021. Epub 2007 Aug 13. PMID 17697704
- [Background] Luijk B, Lindemans CA, Kanters D, van der Heijde R, Bertics P, Lammers JW, Bates ME, Koenderman L. Gradual increase in priming of human eosinophils during extravasation from peripheral blood to the airways in response to allergen challenge. J Allergy Clin Immunol. 2005 May;115(5):997-1003. doi: 10.1016/j.jaci.2005.02.002. PMID 15867857